CLINICAL TRIAL: NCT06122454
Title: A Single-center, Randomized, Open-label, Active-controlled Phase Ic/IIb Study to Evaluate the Efficacy，Safety and Pharmacokinetics of Hepenofovir Fumarate Tablets in Patients With CHB
Brief Title: A Phase Ic/IIb Study to Evaluate the Efficacy，Safety and Pharmacokinetics of HST in Patients With CHB
Acronym: HTS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xi'an Xintong Pharmaceutical Research Co.,Ltd. (Other)
Collaborators: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XAXT-2022-001
Record Dates: First submitted 2023-10-30; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-10

CONDITIONS: Efficacy; Safety; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenofovir alafenamide Fumarate tablets (Active Comparator): TAF is taken orally under postprandial conditions, and subjects begin eating breakfast within 30 minutes of taking the drug. The 25mgQD group is given a single daily dose for 24 consecutive weeks, and continues to take the drug for 48 weeks after completing the 24-week treatment.
  Interventions: Drug: Hepenofovir Fumarate Tablets
- Hepenofovir Fumarate Tablets (Experimental): After taking HTS tablets orally under postprandial conditions, subjects began to eat breakfast within 30 minutes before taking the drug. The 10mgQD and 20mgQD dose groups were administered once daily for 24 consecutive weeks, and continued to be administered for 48 weeks after completing the 24-week treatment. The 40mgQOD group was administered once every other day for 24 weeks, and continued to be administered for 48 weeks after completing the 24-week treatment.
  Interventions: Drug: Hepenofovir Fumarate Tablets

INTERVENTIONS:
Drug: Hepenofovir Fumarate Tablets — Each subject received multiple doses of the test drug/control drug and completed safety, efficacy, and PK evaluations
  Other Names: Tenofovir alafenamide Fumarate tablets

SUMMARY:
The goal of this a clinical trial is to learn about the efficacy，safety and Pharmacokinetics of Hepenofovir Fumarate Tablets（HTS） in patients with CHB. The main questions it aims to answer are：

1. Evaluate the efficacy and safety of multiple doses of continuous administration of HTS in patients with chronic hepatitis B, and compare it with Tenofovir alafenamide Fumarate tablets（TAF）.
2. To evaluate the pharmacokinetic characteristics of HTS in patients with chronic hepatitis B after multiple oral administration.
3. To evaluate the pharmacodynamic changes of HTS in patients with chronic hepatitis B after multiple consecutive administrations, and compare it with TAF.

Positive control drug：Tenofovir alafenamide Fumarate tablets（25mg/d） Test drug：Hepenofovir Fumarate Tablets（10mg/d、20mg/d、40mg/qod） Test process：This study was divided into 4 groups, with the specific list shown below. The initial plan was to include 12 subjects in each group, stratified by HBeAg status, with 4 subjects negative for HBeAg and 8 subjects positive for HBeAg. A total of 48 subjects were included in this trial, and they were randomly assigned to multiple doses at a ratio of 1:1:1:1. The dosing period was 24 weeks. However, after enrolling 37 subjects (29 positive for HBeAg and 8 negative for HBeAg), the protocol was adjusted (V4.0): the remaining 11 subjects would be included, all of whom were over 30 years old with ALT < ULN and met all the inclusion criteria but none of the exclusion criteria. The random assignment was: 7 subjects positive for HBeAg were randomly assigned to HTS 10mg/day, 20mg/day, 40mg/qod and TAF 25mg/day groups at a ratio of 2:2:2:1; and 4 subjects negative for HBeAg were randomly assigned to HTS 10mg/day, 20mg/day, 40mg/qod and TAF 25mg/day groups at a ratio of 1:1:1:1.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily sign the informed consent form.
2. Subjects (including partners) are willing to have no plans for pregnancy from the time of screening to 3 months after the last administration of the study drug and ensure appropriate contraception measures are taken.
3. Male or female subjects (including boundary values) between 18-65 years of age, regardless of gender.
4. Body mass index (BMI) between 18.0-32.0 kg/m2 (including critical values), where BMI = body weight (kg) / height2 (m2).
5. Evidence (including but not limited to outpatient/inpatient medical records/laboratory reports, etc.) to prove a history of positive hepatitis B surface antigen (HBsAg) or positive HBV DNA for at least 6 months at the time of screening, or negative HBcAb IgM and positive HBsAg at the time of screening, or histological examination of liver tissue showing chronic hepatitis B infection.
6. HBeAg-positive patients with HBV DNA ≥ 2.0×104 IU/mL and HBeAg-negative patients with HBV DNA ≥ 2.0×103 IU/mL at the time of screening.
7. Subjects with ALT between 1.2×ULN and 10×ULN within 7 days of screening, or subjects over 30 years of age with ALT less than 1.2×ULN; total bilirubin (TBIL) ≤ 2×ULN;
8. Creatinine clearance rate ≥ 70 mL/min [calculation formula: Ccr: (140-age)×weight (kg) / (0.818×Scr) (μmol/L), female×0.85];
9. Subjects who have not used anti-HBV nucleotide/nucleoside therapy, interferon therapy, or immunomodulators within the previous 6 months prior to screening;
10. Subjects who fully understand the trial process, possible adverse reactions, and can complete the trial according to the protocol plan.

Exclusion Criteria:

1. Subjects with a history of allergies to HTS and TAF, or any other similar drugs, metabolites, or excipients;
2. Subjects who participated in other drug clinical trials within one month prior to the study;
3. Subjects with positive results for hepatitis C antibody, hepatitis C core antigen, HIV antibody, or syphilis antibody screen (if syphilis antibody positive, additional rapid plasma reagin test (RPR) is required, and the investigator should use the results to determine if there is a positive reaction);
4. Subjects with any known disorders in glutathione metabolism (e.g., glutathione deficiency anemia, glutathioneemia), or subjects who require high doses of acetaminophen/Tylenol® (>1 g/day);
5. Subjects with a QTcF interval >470 ms (men) or >480 ms (women) on electrocardiogram at the time of screening (corrected using Fridericia's formula), or any other electrocardiogram abnormalities deemed to be clinically significant by the investigator;
6. Subjects with a history of persistent substance abuse in the past or recent times;
7. People who smoke and drink excessively (14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of hard liquor, or 1 glass of wine; smoking ≥ 5 cigarettes per day);
8. People with decompensated liver disease (Child-Pugh score of B or C), including but not limited to: hepatic encephalopathy, hepatorenal syndrome, variceal bleeding, ascites, or a history of HCC;
9. People with an alpha-fetoprotein (AFP) level > 50 ng/mL at the time of screening, or with imaging suggesting the possibility of malignant liver lesions;
10. People with a history of malignancy within the past 5 years [exceptions: surgically resected and completely cured specific cancers (such as skin basal cell carcinoma or squamous cell carcinoma) or cervical intraepithelial neoplasia];
11. People with a history of organ transplantation or bone marrow transplantation;
12. People who require long-term use of immunosuppressants or drugs with a high risk of liver or kidney toxicity (such as dapsone, erythromycin, fluconazole, ketoconazole, rifampicin, etc.);
13. Pregnant or breastfeeding women or with positive serum pregnancy results;
14. People with other significant liver diseases in addition to hepatitis B, including but not limited to chronic alcoholic hepatitis, drug-induced hepatitis, autoimmune liver disease, etc.
15. Other serious diseases of important organs include but are not limited to definite medical history of nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and skeletal muscle system (such as poorly controlled diabetes (type 1 diabetes or uncontrolled type 2 diabetes (HbA1c≥9.0%)), hypertension that is not well-controlled after medication (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg), etc.), which the investigator believes makes the subject unsuitable for participation in this study;
16. A history of swallowing difficulties or any gastrointestinal diseases that affect drug absorption;
17. Donating blood or losing blood >500 mL within 2 months prior to screening, or donating plasma within 14 days prior to screening;
18. Any significant clinical and laboratory abnormalities (neutrophil count <1.2×109/L during screening; platelet count <80×109/L during screening; hemoglobin <90g/L during screening; international normalized ratio (INR) >1.5 during screening), or investigator believes it affects safety evaluation.
19. Screening urine test: proteinuria > 1+;
20. Positive urine drug screen (morphine, cannabis) or positive breath alcohol test;
21. Subjects who may not be able to complete the trial for other reasons or who the investigator believes should not be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-06-06 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Quantification of HBV DNA | Screening period，week2（Day15±3），week4（Day29±3），week8（Day57±3），week12 （Day85±5），week16（Day113±5），week20（Day141±5），week24（Day169±5），week28（Day197±5）， week32（Day225±5），week36（Day253±5），week40（Day281±5），week44（Day309±5），week48（Day335 QOD or Day336QD ±5）
  HBV DNA
Quantification of HBV markers | Day1 before administration，week12（Day85±5），week24（Day169±5）， week36（Day253±5），week48（Day335 QOD or Day336QD ±5）
  HBsAg ，HBeAg
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | during the intervention、within 4 weeks of completion of treatment
  Symptoms and physical examination, clinical laboratory tests (blood routine, blood biochemistry, coagulation profile, urine routine, thyroid function test), thyroid ultrasound, abdominal ultrasound, vital signs (blood pressure, pulse, respiration and body temperature), 12-lead electrocardiogram, bone density, monitoring and recording of adverse events and concomitant medication.
Area Under the Plasma Concentration Versus Time Curve (AUC) of HTS and TFV | 0min，15min，30min，1hour，1.25hour，1.5hour，2hour，2.5hour，3hour，4hour，5hour，6hour，8hour，12hour，24hour，48hour
  The experimental group measured the concentrations of hepranofovir and tenofovir (TFV), while the control group measured the concentrations of tenofovir (TFV)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Jilin, Changchun, China

IPD SHARING:
Plan to Share IPD: No